CLINICAL TRIAL: NCT00844909
Title: A Phase 1 Study to Evaluate the Pharmacokinetics and Safety of CNTO136 Following a Single Subcutaneous Administration to Healthy Japanese and Caucasian Subjects.
Brief Title: A Study of the Safety and How the Body Effects a Drug CNTO 136 in Healthy Male Japanese and Caucasian Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centocor, Inc. (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: CR015910
Record Dates: First submitted 2009-02-13; First posted 2009-02-16 (Estimated); Last update posted 2010-04-27 (Estimated); Status verified 2009-10

CONDITIONS: Healthy
Keywords: CNTO 136; safety; pharmacokinetics; healthy Japanese; healthy Caucasian; Phase I; antibody; male.
MeSH Terms: interventions — sirukumab

INTERVENTIONS:
Drug: CNTO 136

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and how the body affects the drug CNTO 136 in healthy Japanese and Caucasian volunteers.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, double-blinded study to assess the safety and pharmacokinetics of CNTO 136. In a randomized trial, study medication (CNTO 136 or placebo) is assigned by chance. Double-blinded means that neither the investigator nor the volunteer know which of the study medication they have been assigned to receive. Pharmacokinetics is the study of levels of CNTO 136 circulating in your blood over time. The study population will all be male and consist of 30 Japanese and 30 Caucasian volunteers. Three dose levels of study agent will be assessed. Participants will be required to stay at the research center after study agent administration for the inpatient portion of the study and then required to return for out-patient visits. One of 3 dose levels of CNTO 136 will be given just under the skin (subcutaneous (SC)). The length of this study will be about 20 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Demonstrate an understanding of the study and sign an informed consent form
* Healthy with no clinically relevant abnormalities as determined by medical history, physical examination, blood chemistry assessments, hematologic assessments including complete blood count (CBC), coagulation tests, urinalysis, measurement of vital signs, and ECG
* Japanese volunteers must have been born in Japan, have resided outside of Japan for no more than 5 years, and have Japanese parents and maternal and paternal grandparents. Caucasian subjects must have Caucasian parents
* Have a weight in the range of 60 kg to 90 kg (inclusive), body mass index (BMI) of 19 kg/m2 to 29 kg/m2
* Nonsmoker or agree to smoke no more than 10 cigarettes or 2 cigars per day throughout the study.

Exclusion Criteria:

* Currently have, or have a history of, disease or dysfunction of the pulmonary, cardiovascular, endocrine, hematologic, neurological, immune, gastrointestinal, genitourinary, or other body system, that is clinically significant in the opinion of the investigator
* Have any underlying physical or psychological medical condition that, in the opinion of the investigator, would make it unlikely that the healthy volunteer will complete the study
* Have evidence of any chronic medical condition requiring prescription medications (eg, hypertension, elevated cholesterol/triglycerides, asthma, or diabetes)
* Currently have any known malignancy or have a history of malignancy
* Have had major or traumatic surgery within 12 weeks of screening or any surgery within 1 week.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2009-01; Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of a single SC administration of CNTO 136 in healthy Japanese and Caucasian volunteers

SECONDARY OUTCOMES:
Pharmacokinetics and immunogenicity of a single SC administration of CNTO 136.

CONTACTS AND LOCATIONS:
Overall Officials: Centocor, Inc. Clinical Trial, Study Director — Centocor, Inc.